CLINICAL TRIAL: NCT06456255
Title: Bupivacaine With Epinephrine vs Sham Injections During Endoscopic Sinus Surgery: a Double Blind, Randomized Controlled Trial
Brief Title: Bupivacaine and Epinephrine Injection Study
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Amin Javer (Other)
Responsible Party: Sponsor-Investigator, Amin Javer, Clinical Professor, St. Paul's Hospital, Canada
Organization: St. Paul's Hospital, Canada (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H24-01167
Record Dates: First submitted 2024-05-27; First posted 2024-06-13 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Sinus Disease; Anesthesia; Bleeding
Keywords: endoscopic sinus surgery; bupivacaine; epinephrine
MeSH Terms: conditions — Paranasal Sinus Diseases; Hemorrhage | interventions — Bupivacaine; Epinephrine; salicylhydroxamic acid

STUDY DESIGN:
Intervention Model Description: We propose a double-blind, parallel arm, randomized controlled trial evaluating whether injecting 0.25% bupivacaine with 1:200,000 epinephrine is superior to no injection (sham procedure) during ESS.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Injection (Experimental): - Injection 0.25% bupivacaine with 1:200,000 epinephrine
  Interventions: Drug: Sensorcaine with Epinephrine
- Sham injection (Placebo Comparator): - Sham injection (only puncture, no injecting anything)
  Interventions: Other: Sham injection

INTERVENTIONS:
Drug: Sensorcaine with Epinephrine — The combination contains 0.25% bupivacaine hydrochloride (2.5 mg/mL) and epinephrine bitartrate [(1:200,000) 5 mcg/mL] per vial.
  Arms: Injection
Other: Sham injection — Punctures without any medication injected onto the septum
  Arms: Sham injection

SUMMARY:
Endoscopic sinus surgery (ESS) is a common otolaryngologic procedure that aims to remove the partitions that separate the sinus cavities, remove inflamed tissue, and optimize the sinuses for topical medication use. In this procedure, the surgeon will inject a combination of drugs, local anesthetics, and vasoconstrictors, to reduce bleeding and improve visualization. However, previous studies have shown similar results when injected with only saline. In this study, investigators want to determine if the injection of local anesthesic+vasoconstrictor compared to no injection at all makes any difference in improving the surgeon's visualization during an ESS.

ELIGIBILITY:
Inclusion Criteria:

* Age 19 years or older
* Scheduled for primary ESS (including septoplasty)

Exclusion Criteria:

* Cystic fibrosis
* Systemic vasculitis or any bleeding disorders
* Known or suspected hypersensitivity to bupivacaine or epinephrine
* Previous sinus surgery
* Inhaled drug use (i.e., cocaine) in the preceding 6 months
* Nasal tumors
* Patients on antiarrhythmics.
* Patients with history of severe liver illness.
* Patients identified as high-risk for complications during preoperative assessment with the anesthesiologist (e.g. untreated hypertension, ischemic heart disease, cerebral vascular insufficiency, heart block, peripheral vascular disorder, uncontrolled hyperthyroidism and diabetes)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-11-15 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Boezzart bleeding score | throughout study completion, one day study visit
  Change in mean surgical field quality as determined by the Boezzart bleeding score. Boezaart score of 0 indicates no bleeding, whereas the maximum score of 5 indicates severe bleeding (constant suctioning required).

SECONDARY OUTCOMES:
Total blood loss | throughout study completion, one day study visit
  Change in total blood between injection and sham group measured in millilitres
Surgical time | throughout study completion, one day study visit
  Change in surgical time between injection and sham group measure in minutes
Mean arterial pressure (MAP) | throughout study completion, one day study visit
  Change in Mean arterial pressure (MAP) between injection and sham group measured in millimeters of mercury (mm Hg)
Postoperative bleeding | throughout study completion, one day study visit
  Change in postoperative bleeding between injection and sham group measured in mililiters
Postoperative pain | throughout study completion, one day study visit
  Change in postoperative pain between injection and sham group measured with a Visual Analog Scale (VAS) grading from 0 (no pain) to 5 (severe pain)

CONTACTS AND LOCATIONS:
Locations (1):
- St.Paul's Hospital Sinus Center, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No